CLINICAL TRIAL: NCT03270228
Title: Natural History of Nonspecific Pleuritis Diagnosed After Video-assisted-thoracoscopic-surgery
Status: Completed | Type: Observational
Sponsor: Naestved Hospital (Other)
Responsible Party: Principal Investigator, Simon Reuter, Ph.d.-Student, Naestved Hospital
Other Study IDs: NSP
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Pleural Effusion Due to Another Disorder (Disorder)
Keywords: Incidence of cancer; Survival

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Nonspecific pleuritis after VATS thoracoscopy — Patients with a pleural effusion with unknown origin after a VATS thoracoscopy is classified as nonspecific pleuritis.

SUMMARY:
The investigators want to determine the incidence of malignant disease, type of malignant disease and overall survival in patients diagnosed with NSP after VATS.

DETAILED DESCRIPTION:
Using Landspatientregisteret (LPR) (the National Patient register) the investigators will identify patients who have received a thoracoscopic pleural-biopsy using the SKS-codes KGAC01 and/or KGAA31 and/or KGAC00. From LPR and Cancerregisteret (the National Cancer-register) the investigators will receive diagnosis and additional descriptive data. From dødsårsagsregisteret (the National cause-of-death-register) death date and further descriptive data will be acquired.

Patients with NSP will be identified as patients with no diagnosis six months after pleural-biopsy, despite a thorough investigation.

Patients with a malignant effusion and non-malignant effusion (with known cause) will be used for survival analysis and comparison.

Data Data will be registered in the individual patients CRF (Case Report File) (digital) and will be transferred to a database-program for further processing. Background-variables will be used to describe the study population. Only study-coordinators will have access to data. All data including back-up will be stored and kept in a locked cupboard in a locked room. Only study coordinators possess relevant keys.

Statistics The investigators define significance level (α) as 0.05, and power (β) as 0.80. Descriptive data will be analysed using nonparametric statistics: Chi2-test for categorical data and Mann-Whitney for discrete data. Statistical significance is defined as: p-value < 0.05.

The overall survival of patients with NSP will be analysed using a Caplan-Meier plot and comparison of NSP patients to patients with malignant pleural-effusion the investigators use the Logrank test.

All statistical tests is conducted using STATA14 (4905 Lakeway Dr., College Station, TX 77845).

Ethics This study will not require the approval from Videnskabsetisk komité (the Health Research Ethics Committee), but approval will be sought from Datatilsynet (the Danish Data Protection Agency).

All results will be stored and analysed by computer, and the patients' anonymity will be secured according to the national laws. The data will be stored (anonymised), after completion of the study: data containing cpr.-numbers will be stored behind double-lock at the department.

No patients or investigators have economic incentives for completing the project.

Economy

Expenses related to gathering of data including contact with LPR, Dødsårsagsregisteret and the Danish Cancer Register are already financed through primary investigators PhD-project.

Publication The results from the study will be presented at international scientific congresses and published in international journals. Positive as well as negative results will be published. The scientists right to freely publish the results cannot be limited. All information will be passed anonymously.

The order of authors will follow the Vancouver Declaration, and will thus reflect the amount and significance of work relevant to the specific manuscript.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a VATS thoracoscopy

Exclusion Criteria:

* None

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a VATS thoracoscopy
Sampling Method: Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Incidence of cancer | 10 years
  Percentage

SECONDARY OUTCOMES:
Type of cancer | 10 years
  Lung cancer, mesothelioma etc.
Survival of patients | 10 years
  Comparison of patients with a benign cause, a malignant cause and nonspecific pleuritis

CONTACTS AND LOCATIONS:
Overall Officials: Simon Reuter, MD, PhD, Principal Investigator — Naestved Hospital
Locations (1):
- Naestved Hospital, Næstved, Denmark